CLINICAL TRIAL: NCT04974268
Title: Reduction of Lymphedema Secondary to Breast Cancer Through a Structured Exercise and Weight Loss Program. Randomized Controlled Trial
Brief Title: Reduction of Lymphedema Secondary to Breast Cancer
Acronym: EJERDIETLIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EJERDIETLINF
Record Dates: First submitted 2021-06-23; First posted 2021-07-23 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Lymphedema
Keywords: Lymphedema; breast cancer; strength training; body composition; body mass index; exercise capacity; health-related quality of life; memory; hypocaloric diet; Mediterranean diet
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Weight Reduction Programs

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise and nutritional program (Experimental): Intervention group that receives supervised exercise and weight loss program based on individual and group intervention with Mediterranean diet and substitute for a daily meal (non-mandatory), manual lymphatic drainage and compression garment if there is more than 600 ml of excess volume in the limb affected.
  Interventions: Other: Specific supervised exercise and weight loss program
- Control Group (No Intervention): Control group will receive recommendations for aerobic unsupervised exercise 150 min per week, standard dietary recommendations (Mediterranean diet pattern and 1800 Kcal diet), manual lymphatic drainage and compression garment if there is more than 600 ml of excess volume in the limb affected.

INTERVENTIONS:
Other: Specific supervised exercise and weight loss program — Intervention group that receives supervised exercise and weight loss program based on individual and group intervention with Mediterranean diet and substitute for a daily meal, manual lymphatic drainage and compression garment if there is more than 600 ml of excess volume in the limb affected.
  Arms: Exercise and nutritional program

SUMMARY:
This study evaluates the reduction of lymphedema and its complications in obese women treated with a muscle training and weight loss program as well as the improvement body composition, muscle strength, quality of life and neurocognitive function, compared to a conventional treatment control group.

DETAILED DESCRIPTION:
Introduction: Breast cancer is the most frequent tumour in women. Breast cancer-related lymphedema (BCRL) occurs in 10 to 36% of patients undergoing dissection and emptying of axillary nodes and between 5 and 17% undergoing sentinel node biopsy. BCRL is associated with discomfort, pain, risk of infections, disability, symptoms of depression and anxiety and worse quality of life. The prevalence of persistent lymphedema increases with the presence of obesity.

Aim: In overweight or obese women with BCRL to assess whether a muscle training and weight loss program reduces lymphedema volume and its associated complications, as well as improves body composition, muscle strength, quality of life and neurocognitive function, compared to a conventional treatment control group.

Methodology: Open prospective randomized trial of 2 parallel arms. Subjects: patients referred to the Rehabilitation Unit with lymphedema secondary to breast cancer and overweight or obesity. The control group will receive the usual treatment and general dietary recommendations and the intervention group will carry out a program of supervised exercise (strength and aerobic) and weight loss (based on the Mediterranean diet and with a meal replacement). The change in volume in the limb affected by lymphedema, segmental body composition and phase angle (impedance measurement), muscular strength (hand dynamometry), level of physical activity (IPAQ), dietary parameters, quality of life (FACB+4) will be assessed. Cognitive function (Memory FSRCT test), psychological symptoms (anxiety and depression by means of HADS) NS biochemical parameters (albumin, prealbumin, lipids, CRP, 25-OH vitamin D and insulin) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years and under 80 who have lymphedema diagnosed according to the truncated cone formula (increase of > 200 ml with respect to the contralateral) and are referred to Rehabilitation for treatment.
* Having completed the chemotherapy and radiotherapy treatment at least 6 months prior to randomization.
* Not having received manual lymphatic drainage in the 2 months prior to the intervention.
* BMI > 25 y < 40 kg/m2.
* Signature of informed consent.

Exclusion Criteria:

* Traumatological, neurological, rheumatological or cardiovascular problems that prevent patients from performing the training.
* Phase IIIB structured lymphedema
* Metastatic disease.
* Illness that prevents the subject from carrying out the program.
* Unstable heart disease
* Ejection fraction of the left ventricle higher than 35.
* Voluntary or involuntary weight loss > 10% in the last 3 months.
* Illiterate.
* Those who do not sign the informed consent to participate in the study.
* Abusive intake of alcohol or other dependencies that in the opinion of the investigator could interfere with the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
To assess the change in volume in the limb affected by lymphedema in the intervention group vs control. | Baseline, 3rd and 6th month visits
  It will be studied whether a reduction of 200 ml of the affected arm is achieved with respect to itself and / or with respect to the healthy one, after training.

SECONDARY OUTCOMES:
BMI (body mass index) changes | Baseline, 3rd and 6th month visits
  Measured by body composition analysis
Change in weight | Baseline, 3rd and 6th month visits
  Weight in kg
Change in fat free body mass | Baseline, 3rd and 6th month visits
  Fat free body mass in kg assessed by bioelectrical impedance analysis
Change in total fat mass | Baseline, 3rd and 6th month visits
  Total fat mass in kg
Change in water on arm affected by lymphedema | Baseline, 3rd and 6th month visits
  Water in ml
Change in water on arm not affected by lymphedema | Baseline, 3rd and 6th month visits
  Water in ml
Peripheral muscle strength | Baseline, 3rd and 6th month visits
  Measured by hand and quadriceps dynamometry. Assess if strength improves after training.
Level of physical activity (IPAQ questionnaire) | Baseline, 3rd and 6th month visits
  Assess whether the level of physical activity improves after training and motivation sessions.
Quality of life (through the FACB + 4 test) | Baseline, 3rd and 6th month visits
  Assess if it improves after training and at 6 months of follow-up.
Change in serum albumin concentration | Baseline, 3rd and 6th month visits
  Serum albumin in g/dl
Change in serum prealbumin concentration | Baseline, 3rd and 6th month visits
  Serum prealbumin in mg/dl
Change in cholesterol concentration | Baseline, 3rd and 6th month visits
  Serum cholesterol in mg/dl
Change in LDL concentration | Baseline, 3rd and 6th month visits
  Serum LDL in mg/dl
Change in TG concentration | Baseline, 3rd and 6th month visits
  Serum TG in mg/dl
Changes in plasma levels of high sensitivity C reactive protein (hs-CRP) | Baseline, 3rd and 6th month visits
  Plasma levels of high sensitivity C reactive protein (hs-CRP) in mg/dl
Changes in metabolic control | Baseline, 3rd and 6th month visits
  Measured as HbA1c (glycated hemoglobin)
Changes in insuline resistance | Baseline, 3rd and 6th month visits
  Measured aas HOMA-IR (homeostatic model assessment of insulin resistance)
Changes in vitamin D | Baseline, 3rd and 6th month visits
  Serum vitamin D in ng/ml
Diet composition | Baseline, 3rd and 6th month visits
  Adherence to the Predimed Plus diet pattern 17 (0 - minimum adherence, 17 - maximum adherence)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Olveira, MD, PhD, Principal Investigator — Hospital Regional Universitario de Málaga - FIMABIS
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Málaga, Spain